CLINICAL TRIAL: NCT01582334
Title: Easypod Connect: A National, Multicentre, Observational Registry to Evaluate Adherence and Long Term Outcomes of Therapy in Paediatric Subjects Using "Easypod™" Electromechanical Device for Growth Hormone Treatment in Argentina
Brief Title: To Assess the Level of Adherence of Subjects Receiving SAIZEN® Via Easypod™ in Argentina
Acronym: ECOS ARG
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Quimica Argentina S.A.I.C (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200104-532
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Growth Disorders
Keywords: Growth disorders; Saizen; Easypod; Growth hormone; Pediatric subject
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: easypod™ — Saizen (Somatropin) as per Summary of Product Characteristics administered by easypod™
  Other Names: Somatropin

SUMMARY:
This is an Argentinian, Multicentre, Observational Study to evaluate Adherence and Long Term Outcomes of Therapy in paediatric subjects using easypod™ electromechanical device for growth hormone treatment and to assess the level of adherence of subject receiving SAIZEN® via easypod™.

DETAILED DESCRIPTION:
Subjects will be enrolled in a multicenter longitudinal observational study. Parents/subjects will provide their Informed Consent/assent to upload their data for population-based analyses and, ultimately, clinical outcomes. Adherence data will be primarily derived from the easypod™ device combined with physician data entry of outcome measures. Data will be collected both retrospectively and prospectively. This will allow the establishment of adherence profiles and explore the hypothesis that patient adherence support programs improve adherence and subsequent clinical outcomes. Collected data will be also analyzed in a multinational pooled analysis of comparable national studies.

Primary Objective:

• To assess the level of adherence of subjects receiving SAIZEN® via easypod™

Secondary Objectives:

* To describe the impact of adherence on clinical outcomes for subject receiving SAIZEN® via easypod™
* To identify adherence subject profiling
* To assess the impact of adherence on Insulin-like Growth Factor 1 (IGF1) (i.e. above, below or within normal ranges)

ELIGIBILITY:
Inclusion Criteria:

* Administered growth hormone via the easypod™ electromechanical device according to Summary of Product Characteristic (SmPC)
* Over the age of >2 years
* Under <18 years of age, or over 18 without fusion of growth plates
* Parent's or guardian's written informed consent, given before entering data into the observational study, with the understanding that the subject or parent/guardian may withdraw consent at any time without prejudice to future medical care. If the child is old enough to read and write, a separate assent form will be given as defined in the appropriate jurisdiction of each country

Exclusion Criteria:

* Subjects taking growth hormone in whom growth plates have fused (i.e. for taking growth hormone for it's metabolic effects)
* Contra-indications to SAIZEN® as defined in the SmPC
* Use of an investigational drug or participation in another interventional clinical study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric subjects (aged 2-18) who are taking SAIZEN® for registered indications using the easypod™ electromechanical device.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-03-31 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Mean percent of daily recorded adherence | At least 6 months and up to 5 years

SECONDARY OUTCOMES:
Correlation of adherence and growth outcome after each year of SAIZEN® treatment with easypod™ | At least 6 months and up to 5 years
  Correlation of adherence and growth outcome (change in: height velocity (HV), height velocity-standard deviation score (HV-SDS), height, height-standard deviation score(height SDS)) after each year of SAIZEN® treatment with easypod™
Subject adherence profile based on age, gender, indication, self-injection or not, time on treatment | At least 6 months and up to 5 years
Correlation of adherence with current IGF-1 status (i.e. above, below or within normal ranges) | At least 6 months and up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Quimica Argentina S.A.I.C
Locations (1):
- For Recruiting Locations in Argentina, Please Contact the Merck KGaA Communication Center, Argentina

REFERENCES:
- [Result] Koledova, E. et al. (2017) Analysis of results from the global, 5-year Easypod™ Connect Observational Study (ECOS) study in children with growth disorders. 10th International Meeting for Pediatric Endocrinology; 2017 Sep 14-17; Washington, DC.
- [Result] Wit, JM. et al. (2017) Effect of adherence on the 2-year growth response to growth hormone treatment in prepubertal children with idiopathic isolated growth hormone deficiency participating in the EasypodTM Connect Observational Study (ECOS). 10th International Meeting of Paediatric Endocrinology; 2017 Sep 14-17; Washington, DC.